CLINICAL TRIAL: NCT05278546
Title: A Phase Ia, Multicenter, Open-label Study of ILB2109 in Patients With Advanced Solid Malignancies
Brief Title: A Study of ILB2109 in Patients With Advanced Solid Malignancies
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Innolake Biopharm (Industry)
Collaborators: Shanghai East Hospital (Other); Shandong Cancer Hospital and Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CILB2109A101
Record Dates: First submitted 2022-02-23; First posted 2022-03-14 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment Arm (Experimental): There are nine escalating dose cohorts.
  Interventions: Drug: ILB2109

INTERVENTIONS:
Drug: ILB2109 — ILB2109 tablets by mouth once per day at dosages prespecified by the protocol. Participants will continue treatment until the end of the study in the absence of unacceptable toxicities and confirmed disease progression.

SUMMARY:
This is a multicenter, open-label, phase Ia study to evaluate the safety, tolerability and preliminary efficacy of ILB2109, a A2a receptor antagonist, in patients with locally advanced or metastatic solid malignancies.

DETAILED DESCRIPTION:
This is a two-part study consists of dose escalation and dose expansion. The dose escalation part adopts a 3+3 protocol design and consists of 5 cohorts. Based on the data obtained from the escalation study, selected cohorts will be expanded to further investigate the safety and efficacy of the study drug. The escalation part consists of a single-dose cycle (Cycle 0) followed by multiple-dose cycles (Cycle 1 and above). Subjects will be assessed for safety and efficacy outcomes at pre-specified time points.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytological confirmed, solid, malignant tumor that is refractory to standard therapy or for which no standard of care regimen currently exists;
* At least one assessable tumor lesion according to RECIST v1.1 in dose escalation part of the study ; At least one measurable tumor lesion according to RECIST v1.1 in dose expansion part of the study;
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1;
* Major organ functions are normal, meets pre-specified lab requirements;
* Females of reproductive age must have a negative serological hCG test during the screening period;
* Subjects of reproductive age (both male and female) must agree to use contraceptive methods from signing Informed Consent to 90 days post the last dose;

Exclusion Criteria:

* Has received any investigational medicinal product or other systemic anticancer treatment within 4 weeks prior to the first dose of study treatment;
* Unable to take medication orally, or has impaired GI function;
* Has received systemic glucocorticoids (prednisone>10 mg/ day or an equivalent dose of another drug of the same class) or other immunosuppressants within 14 days prior to the first dose of study treatment;
* Has received live, attenuated vaccines within 4 weeks prior to the first dose of study treatment;
* Has active infection that requires intravenous anti-infective therapy;
* History of HIV infection, or other acquired, congenital immunodeficiency disease, or a history of organ transplantation;
* History of serious cardiovascular and cerebrovascular diseases;
* History of adverse effect from previous antineoplastic therapy that has not returned to CTCAE grade 5.0 ≤1;
* Cerebral parenchymal or meningeal metastasis;
* History of ≥ Grade 3 irAE or ≥ Grade 2 myocarditis from previous immune therapy;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-04-11 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
The Incidence of DLTs | At the end of Cycle 0 and 1 (Cycle 0 is 3 days, Cycle 1 is 21 days)
  The incidence rate of Dose Limiting Toxicities (DLTs)
MTD | 30 Months
  Determining the maximum tolerated dose (MTD) for subsequent studies
RD | 30 Months
  Determining the Recommended Dose (RD) for subsequent studies

SECONDARY OUTCOMES:
Safety Outcomes | From Informed Consent to 28 days after the last dose, expected follow-up period 6 months
  Determining the incidence rate, type and severity of Treatment Emergent Adverse Event (TEAE), Treatment Emergent Serious Adverse Event (TESAE), and lab abnormalities (hematology and major organ function lab tests) based on NCI-CTCAE 5.0;
Objective Response Rate (ORR) | Tumor assessment every 6 weeks (+/- 7 days) until disease progression, expected follow-up period 6 months
  n tumor treatment, the proportion of patients whose tumor volume has shrunk to a predetermined value and can be maintained for a certain period of time. It includes the proportion of patients with complete remission (CR) and partial remission (PR) to the total number of evaluable cases.
Progression Free Survival (PFS) | Tumor assessment every 6 weeks (+/- 7 days) until disease progression, expected follow-up period 6 months
  The time from randomization of patients to the onset of disease progression.
Overall Survival (OS) | Tumor assessment every 6 weeks (+/- 7 days) until disease progression, expected follow-up period 6 months
  The time from randomization to death for any reason
1-Year OS | Tumor assessment every 6 weeks (+/- 7 days) until disease progression, expected follow-up period 6 months
  The probability of a survival time of 1 year after treatment for this disease
Time To Response (TTR) | Tumor assessment every 6 weeks (+/- 7 days) until disease progression, expected follow-up period 6 months
  Time from the start of treatment to the first objective tumor response
Duration Of Response (DOR) | Tumor assessment every 6 weeks (+/- 7 days) until disease progression, expected follow-up period 6 months
  The time from response to progression/death
Clinical Benefit Response (CBR) | Tumor assessment every 6 weeks (+/- 7 days) until disease progression, expected follow-up period 6 months
  The total percentage of patients who achieved a complete response, partial response, or had stable disease for 6 months or more.
Maximum Plasma Concentration (Cmax) | Blood samples will be collected at pre-specified time points in Cycles 0, 1 and 2 (Cycle 0 is 3 days, Cycles 1&2 each is 21 days)
  Characterize the single-dose and multiple-dose plasma concentration of ILB2109
Area Under the plasma drug concentration-time Curve (AUC) | Blood samples will be collected at pre-specified time points in Cycles 0, 1 and 2 (Cycle 0 is 3 days, Cycles 1&2 each is 21 days)
  Characterize the single-dose and multiple-dose plasma concentration of ILB2109

OTHER OUTCOMES:
Plasma Concentration of Downstream Signaling Protein | Blood samples will be collected at pre-specified time points in Cycles 0 and 1 (Cycle 0 is 3 days, Cycle 1 is 21 days)
  Characterize the relationship between the plasma concentration of ILB2109 and the level of a downstream signaling protein to evaluate the pharmacodynamics of ILB2109.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, M.D., Principal Investigator — Shanghai East Hospital
Locations (2):
- China (2):
  - Shandong Cancer Hospital and Institute, Jinan, Shandong
  - Shanghai East Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No